CLINICAL TRIAL: NCT00248443
Title: Severe Acute Respiratory Failure in Hematology and Cancer Patients Without Bronchoalveolar Lavage. A Multicentric Randomized Controlled Trial
Brief Title: Réa-MiniMax: Severe Acute Respiratory Failure in Hematology and Cancer Patients Without Bronchoalveolar Lavage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Saliha DJANE, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P040424
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2007-03

CONDITIONS: Lymphoma; Cancer; Acute Respiratory Failure; Leukemia
Keywords: Haematology and cancer patients; Acute respiratory failure; Bronchoalveolar lavage; Non invasive diagnostic tools; Mechanical ventilation; Intensive Care
MeSH Terms: conditions — Lymphoma; Neoplasms; Leukemia | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Fiberoptic bronchoscopy and bronchoalveolar lavage

SUMMARY:
The MiniMax® study is a multicenter randomized controlled study aimed at demonstrating that a combination of non-invasive diagnostic tools are as effective as fiberoptic bronchoscopy and bronchoalveolar lavage (FO-BAL) in performing the etiological diagnosis of acute respiratory failure in cancer patients.

DETAILED DESCRIPTION:
Acute respiratory failure is a dreadful complication in cancer patients. Indeed, about 20% of the patients will present with pulmonary infiltrates, but Intensive Care Unit (ICU) admission and mechanical ventilation will be needed in half of them resulting in mortality for most of the patients. Managing cancer patients with respiratory failure implicates three mandatory tasks: 1) early antibiotics administration covering suspected pathogens; 2) search for the actual aetiology; and 3) adequate supportive care with access to invasive or non invasive respiratory support. Performing the etiological diagnosis is crucial. Fiberoptic bronchoscopy and bronchoalveolar lavage (FO-BAL) remains the cornerstone of the management of pulmonary infiltrates in cancer patients. However, non-invasive diagnostic tools have been validated in the recent years. Diagnostic and therapeutic impacts of FO-BAL are only of 30% to 60% and 15% to 60% respectively. In neutropenic patients and recipients of bone marrow or stem cell transplantation, this impact is significantly altered. Moreover, reports have highlighted significant rates of complications such as haemorrhage (5%), respiratory deterioration (11% to 40%), possibly heading to intubation and subsequent death. Therefore, balancing advantages to risks of FO-BAL is in order. The MiniMax® study is a multicenter randomized controlled study aimed at demonstrating that a combination of non-invasive diagnostic tools are as effective as FO-BAL in performing the etiological diagnosis of acute respiratory failure in cancer patients. In addition, these non-invasive tests might not lead to deterioration of the respiratory status and corresponding requirement to intubation and mechanical ventilation. The group of investigators is used to manage cancer patients with pulmonary involvement. In the 21 centres, patients will be randomized to be managed either with FO-BAL or with only non-invasive tools. In each case, patients will be managed with the best supportive care including adequate antibiotics, respiratory support and all needed life sustaining therapies. Our hypothesis is to reduce intubation rate using a non-invasive approach (without FO-LBA). Surrogate markers will be hospital mortality and the number of diagnostic procedures in each group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a malignant haemopathy or a cancer
* Patients with severe acute respiratory failure requiring admission to an ICU
* No argument for a congestive cardiac insufficiency (heart failure)
* Patients who provided their informed consent

Exclusion Criteria:

* Age less than 18
* Patient who refuses to undergo fiberoptic bronchoscopy
* Therapeutic limitation
* Patients intubated at ICU admission
* Etiological diagnosis of the acute respiratory failure known
* Lack of available bronchoscopy
* AIDS
* Post-operative direct admission
* Inclusion in another research protocol in the ICU (HURRIET law)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2005-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Reduction in intubation rate | 28 days

SECONDARY OUTCOMES:
Mortality at 28 days | 28 days
Hospital mortality | 28 days
Duration of mechanical ventilation (invasive or non invasive) | 28 days
Psychological aftereffects | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Elie Azoulay, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Réanimation Médicale de l'Hôpital Saint-Louis, Paris, France

REFERENCES:
- [Background] Dunagan DP, Baker AM, Hurd DD, Haponik EF. Bronchoscopic evaluation of pulmonary infiltrates following bone marrow transplantation. Chest. 1997 Jan;111(1):135-41. doi: 10.1378/chest.111.1.135. PMID 8996007
- [Background] White P, Bonacum JT, Miller CB. Utility of fiberoptic bronchoscopy in bone marrow transplant patients. Bone Marrow Transplant. 1997 Oct;20(8):681-7. doi: 10.1038/sj.bmt.1700957. PMID 9383232
- [Background] Murray PV, O'Brien ME, Padhani AR, Powles R, Cunningham D, Jeanes A, Ashley S. Use of first line bronchoalveolar lavage in the immunosuppressed oncology patient. Bone Marrow Transplant. 2001 May;27(9):967-71. doi: 10.1038/sj.bmt.1703020. PMID 11436107
- [Derived] Azoulay E, Mokart D, Lambert J, Lemiale V, Rabbat A, Kouatchet A, Vincent F, Gruson D, Bruneel F, Epinette-Branche G, Lafabrie A, Hamidfar-Roy R, Cracco C, Renard B, Tonnelier JM, Blot F, Chevret S, Schlemmer B. Diagnostic strategy for hematology and oncology patients with acute respiratory failure: randomized controlled trial. Am J Respir Crit Care Med. 2010 Oct 15;182(8):1038-46. doi: 10.1164/rccm.201001-0018OC. Epub 2010 Jun 25. PMID 20581167